CLINICAL TRIAL: NCT03364686
Title: Transfusion of Biotin-Labeled Red Blood Cells for the Evaluation of Genetic Factors That Contribute to Donor Differences in Red Blood Cell Storage and Post-Transfusion Red Blood Cell Recovery
Brief Title: Transfusion of Biotin-Labeled Red Blood Cells
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to enrollment challenges related to COVID and lack of coordinator support
Sponsor: Gladwin, Mark, MD (Individual)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Darrell Triulzi MD, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY19020356; 5R01HL098032-09 (NIH)
Record Dates: First submitted 2017-11-22; First posted 2017-12-06 (Actual); Results first posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-03

CONDITIONS: Healthy Volunteers
Keywords: BioRBCs; Biotin labeled red blood cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Biotin-Labeled Red Blood Cells Infusion (Experimental): Each participant will receive 2 transfusions of biotin labeled red blood cells.
  Interventions: Biological: Biotin-Labeled Red Blood Cells

INTERVENTIONS:
Biological: Biotin-Labeled Red Blood Cells — We will collect 500 mL of blood. The blood will be processed and split into two bags and labeled with a naturally occurring vitamin, biotin. The blood will then be re-infused back into the same participant at 2 time points (5-7 days and 35-42 days after storage).

SUMMARY:
The purpose of this research is to evaluate the impact of genetic and biologic factors in blood donors on red blood cell storage stability after autologous transfusion over the different range of storage period of 5-7 days and 35-42 days in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 years and older
* Weight ≥110 lbs
* Hemoglobin ≥ 12.5 g/dL or hematocrit ≥ 38% for women and hemoglobin ≥ 13.0 g/dL or hematocrit ≥ 39% for men.
* Meet criteria for autologous blood donation

Exclusion Criteria:

* Subjects with a past medical history or symptoms of blood dyscrasia, diabetes mellitus, hyperlipidemia, obstructive sleep apnea, renal disease, congestive heart failure, significant cardiac disease and / or known peripheral arterial disease.
* Moderate to severe systemic hypertension (systolic blood pressure >140 mmHg and/or diastolic blood pressure > 95 mmHg
* Systolic blood pressure <100 mmHg and/or diastolic blood pressure < 60 mmHg on the study day.
* Positive Direct Antiglobulin Test
* Consumption of biotin supplements or raw eggs within 30 days
* Treatment with antibiotics in the week before initiating study participation to avoid suppression of erythropoiesis, which may accompany infection.
* Blood loss in the previous 8 weeks due to epistaxis, trauma, hemoptysis, gastrointestinal bleeding, diagnostic phlebotomy (> 30 ml)
* Subjects who report tobacco or marijuana smoking within 6 months of study.
* Cognitively impaired subjects, or institutionalized persons and subjects unable or unwilling to complete written informed consent
* Subjects with a history of blood donation within the last 56 days.
* Use of other investigational drugs/devices within 30 days of screening.
* Subjects taking any medication for the treatment of diabetes including insulin
* Females of childbearing potential who are pregnant or unwilling to undergo pregnancy testing; females with positive pregnancy testing on screening day will be excluded.
* History of prior transfusion reaction to blood products.
* Allergic reaction to biotin
* Donors with naturally occurring antibodies against BioRBCs will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darrell Triulzi, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Biotin-Labeled Red Blood Cells Infusion
Started | 6
Completed | 4
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Biotin-Labeled Red Blood Cells Infusion
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Biotin Labeled Red Blood Cells
Description: This will be determined using enumeration of biotinylated red blood cells obtained by flow cytometry from blood samples obtained at various time points from subjects with specified genetic mutations, compared with control subjects without the specified mutation. Percentage of Biotin Labeled Red Blood Cells is determined by Biotin Labeled Red Blood Cells in circulation at each time point/baseline Biotin Labeled Red Blood Cells in circulation x 100.
Time Frame: 24 hours, 30 days and 60 days after transfusion
Population: The blood sample at 24 hours from one of the 4 completed subjects was not collected.
Measure: Mean (95% Confidence Interval); unit: percentage of biotin labeled RBC
Arm/Group | Biotin-Labeled Red Blood Cells Infusion
Number analyzed (Participants) | 3
percentage of biotin labeled RBC
  Percentage of Fresh Biotin Labeled Red Blood Cells at 24 Hours | 99.2 [99.2 to 99.3]
  Percentage of Fresh Biotin Labeled Red Blood Cells at Day 30 | 77.2 [74.7 to 79.6]
  Percentage of Fresh Biotin Labeled Red Blood Cells at Day 60 | 54.3 [49.5 to 59.2]
  Percentage of Aged Biotin Labeled Red Blood Cells at 24 Hours | 99.2 [99.1 to 99.3]
  Percentage of Aged Biotin Labeled Red Blood Cells at Day 30 | 75.9 [72.9 to 78.9]
  Percentage of Aged Biotin Labeled Red Blood Cells at Day 60 | 51.9 [45.9 to 57.8]

2. Secondary Outcome: The Percentage of Storage Hemolysis
Description: This will be quantified as percent hemolysis, which accounts for the levels of RBC-derived free hemoglobin in response to cold storage. We will define the associations between the primary endpoints and the quantification of storage hemolysis. Quantification of storage hemolysis is based on this equation: (sample hematocrit x levels of free hemoglobin obtained after centrifugation measured in the supernatant / the total amount of sample hemoglobin before centrifugation) x 100.
Time Frame: 5-7 days and 35-42 days following blood donation
Measure: Mean (Standard Deviation); unit: percentage of storage hemolysis
Arm/Group | Biotin-Labeled Red Blood Cells Infusion
Number analyzed (Participants) | 4
percentage of storage hemolysis
  5-7 days | 0.27 (0.09)
  35-42 days | 0.21 (0.14)

3. Secondary Outcome: The Percentage of Red Blood Cell Osmotic Hemolysis
Description: This will be quantified by the evaluation of osmotic stress assays. We will define the associations between the primary endpoints and the quantification of osmotic hemolysis. The percent osmotic hemolysis is determined by this equation: (supernatant cell-free hemoglobin of pink test-treated RBCs / total amount of hemoglobin) x 100.
Time Frame: 5-7 days and 35-42 days following blood donation
Measure: Mean (Standard Deviation); unit: percentage of osmotic hemolysis
Arm/Group | Biotin-Labeled Red Blood Cells Infusion
Number analyzed (Participants) | 4
percentage of osmotic hemolysis
  5-7 days | 7.4 (4.66)
  35-42 days | 7.9 (6.86)

4. Secondary Outcome: The Percentage of Red Blood Cell Oxidative Hemolysis
Description: This will be quantified by the evaluation of oxidative stress assays. We will define the associations between the primary endpoints and the quantification of oxidative hemolysis. The percent osmotic hemolysis is determined by this equation: (supernatant cell-free hemoglobin of 2,2'-azobis-2-methyl-propanimidamide, dihydrochloride treated RBCs - supernatant cell-free hemoglobin of untreated red blood cells / total amount of hemoglobin) x 100.
Time Frame: 5-7 days and 35-42 days following blood donation
Measure: Mean (Standard Deviation); unit: percentage of oxidative hemolysis
Arm/Group | Biotin-Labeled Red Blood Cells Infusion
Number analyzed (Participants) | 4
percentage of oxidative hemolysis
  5-7 days | 39.93 (12.45)
  35-42 days | 46.90 (21.92)

5. Post Hoc Outcome: Length of Time Biotin-labeled Red Blood Cells Can be Detected Following Infusion
Description: This will be determined using enumeration of biotinylated red blood cells obtained by flow cytometry from blood samples obtained at various time points from subjects.
Time Frame: up to 165 days
Population: The fresh stored blood sample from one participant was not collected and analyzed.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Biotin-Labeled Red Blood Cells Infusion
Number analyzed (Participants) | 4
days
  Fresh Stored Cells: number analyzed (Participants) | 3
  Fresh Stored Cells | 135 (12)
  Stored Cells | 104 (12)

ADVERSE EVENTS:
Time Frame: Day 125-150 post blood transfusion
Arm/Group | Biotin-Labeled Red Blood Cells Infusion
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biotin-Labeled Red Blood Cells Infusion (N=6)
Weakly positive antibodies (Blood and lymphatic system disorders) | 1 (1) — Subject developed transient antibiotin antibodies without evidence of hemolysis. The test was weakly positive at Visit 8 and was undetected at Visit 10.

LIMITATIONS AND CAVEATS:
The clinical trial was terminated early due to challenges with enrollment and lack of study coordinator support. Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/86/NCT03364686/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/86/NCT03364686/ICF_001.pdf